CLINICAL TRIAL: NCT06410846
Title: Feasibility and Effectiveness of a Novel Neck Training Device: A Pilot Study
Brief Title: Feasibility and Effectiveness of a Novel Neck Training Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Landstuhl Regional Medical Center (U.S. Federal Agency)
Collaborators: TriService Nursing Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FY22-03
Record Dates: First submitted 2024-04-15; First posted 2024-05-13 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Injury Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TopSpin device (Experimental): TopSpin360 device/neck strengthening exercises.
  Interventions: Device: TopSpin360
- Control group (Active Comparator): Neck Strengthening exercises.
  Interventions: Other: Neck Strengthening Exercise Plan

INTERVENTIONS:
Device: TopSpin360 — Neck strength and conditioning device used during neck strengthening program.
  Arms: TopSpin device
Other: Neck Strengthening Exercise Plan — Physical therapist designed neck strengthening program.
  Arms: Control group

SUMMARY:
Functional training focusing on dynamic, multiplanar eccentric loading of the neck's complex musculature may provide a unique training effect that may protect against neck injuries and mTBI. The purpose of this study is to test the efficacy and adherence of a 12-week TopSpin360 training regimen on important physiologic and performance outcome measures between an intervention group and a control group. The specific aims are 1) to compare differences in four physiologic neck measures and two TopSpin360 performance measures by group and gender, and 2) to evaluate program adherence.

DETAILED DESCRIPTION:
The study will employ a randomized controlled clinical trial design with pre-and post-exposure testing and comparison of intervention and control groups. Inclusion criteria are active-duty men and women of any rank assigned to LRMC, ages 18-35, own a personal cellphone to download the TopSpin360 App (intervention group), able to attend the two times per week training, and have sufficient time on stations to complete the entire study including post-study measures. Exclusion criteria include any medical profile that prevents full participation in the ACFT, any chronic inner ear abnormalities or history of invasive neck procedures or any gross cervical abnormalities when examined by the staff physical therapist.

Study participants in both groups will be measured at baseline and study conclusion. The intervention will use the TopSpin360 device, and the control group will perform a physical therapist designed neck strengthening program. A certified athletic trainer or physical therapist will lead the intervention group for the 12-weeks duration. Data collected will include demographics, physiologic and performance measures, and program adherence.

ELIGIBILITY:
Inclusion Criteria:

* Healthy active-duty service members of any military rank assigned to LRMC
* 18-35 years old
* assigned to Landstuhl Regional Medical Center
* own a personal cellphone to download the TopSpin360 App (intervention group)
* able to attend the two times per week training
* have sufficient time on station to complete entire study including post-study measures.

Exclusion Criteria:

* any medical profile that prevents full participation in the ACFT
* any chronic inner ear abnormalities (e.g., Meniere's disease or benign positional vertigo)
* history of invasive neck procedures (cortisone injections or neck surgery)
* any known cervical spine disorders (e.g., degenerative changes of the cervical spine) or gross cervical spine abnormalities when examined by the staff physical therapist
* non-US military personnel, i.e., German or Netherlands military personnel etc.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in neck circumference measurement over time | Day 1 and post 12 week exercise follow up visit day
  Describe change in neck measurement (inches) between intervention and control groups and gender. Examiner will use Gulick tape measure at the midcervical spine level at mid-point between the suboccipital junction and the C7 spinous process.
Change in cervical spine range of motion (ROM) measurements over time | Day 1 and post 12 week exercise follow up visit day
  ROM will be measured using smartphone inclinometer and compass measurements of cervical uniplanar (FL/EXT) and multiplanar (rotation) motion .These measurements have been found to be both reliable and 51 valid by Guidetti et.al. (2017) who demonstrated ICC > .99 with minimally detectable change (MDC) of 4-8 degrees and percentage errors between 1-3%.The 52 overcomes the limitation of protractor measurement as a source of error in cervical spine measures as there is no reference to vertical or horizontal, relying on the visual perceptual skills of the examiner and a lack of a standard position.
Change in Maximum Voluntary Isometric Contraction Testing (MVIC) over time | Day 1 and post 12 week exercise follow up visit day
  The hand-held strain gage dynamometer (Lafayette Instruments HHD) will be conducted by the examiner and record the average of 3 trials most representative of best effort. HHD has demonstrated ICCs of .95 between HHD and the gold standard of MVIC measurement using a Cybex isokinetic device in stroke patients and that the make test demonstrated break force ICCs of .981.53 Isokinetic devices (Kin Com and Cybex) and the strain-gage HHD demonstrate a high test-retest reliability (ICC = 0.998) against a known load. MVIC 54 testing using a HHD requires that the examiner elicit the subject's maximum force against the dynamometer and examiner who holds the dynamometer steady. The Lafayette handheld dynamometer utilizes a microprocessor control unit that measures peak force, time to reach peak force, and total test time with an audible tone to indicate the end of preset time. The unit also provides a built-in calibration routine with an internal accuracy of + 1%.
Change in speed for Peak Revolutions per minute (RPM) over time (TopSpin group only) | Day 1 and post 12 week exercise follow up visit day
  An Inflatable pressure biofeedback device is used for the Craniocervical flexion test (CCFT). The CCFT of the deep cervical spine flexors (longus capitus and colli) assesses the activation and isometric endurance of the deep cervical flexors as well as their interaction with the superficial flexors (sternocleidomastoid and anterior scalenes) during five progressive stages of craniocervical flexion, demonstrated 56-58 SCM and AS muscle fatigue during sustained cervical flexion contractions at 25 and 50% of maximum voluntary isometric contraction. Testing will be conducted according to Jull et. al.'s (2008) progressive protocol using a pressure biofeedback device (Figure 5). The CCFT has demonstrated nearly perfect intra-rater (ICC =.98; CI = .99) and inter-rater reliability (ICC = .91). Changes in speed over exercise program will be described.
Change in speed for completion of 60 revolutions over time (TopSpin group only) | Day 1 and post 12 week exercise follow up visit day
  Measure and describe completion of a total of 60 revolutions (30 clockwise and 30 counterclockwise) as quickly as possible. During the test, when the participant completes the first 30 revolutions, they will stop the lever arm in front of their face and then perform the remaining 30 revolutions counterclockwise. The total time is recorded in seconds and is downloaded from the TopSpin app.

CONTACTS AND LOCATIONS:
Overall Officials: William Brown, PhD, Study Director — Martin Army Community Hospital
Locations (1):
- Landstuhl Regional Medical Center, Landstuhl, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No